CLINICAL TRIAL: NCT06640634
Title: Effect of Anodal Transcranial Direct Current Stimulation on Postdural Puncture Headache: Results of Two Randomized Sham - Controlled Trials
Brief Title: Effect of Anodal Transcranial Direct Current Stimulation on Postdural Puncture Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Diego Centonze, Head of Neurology Unit, Neuromed IRCCS
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: PDPH-tDCS
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-10

CONDITIONS: Postdural Puncture Headache; Lumbar Puncture
Keywords: headache; post-dural puncture headache; transcranial direct current stimulation; noninvasive brain stimulation; neuromodulation
MeSH Terms: conditions — Post-Dural Puncture Headache; Headache

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- therapeutic a-tDCS (Th-tDCS) (Experimental): In patients diagnosed with PDPH, three consecutive days of active a-tDCS intervention are performed starting from the day of diagnosis.
  Interventions: Device: active in therapeutic tDCS (Th-tDCS): anodal transcranial Direct Current Stimulation (a-tDCS)
- sham in therapeutic t-DCS (Th-tDCS) (Sham Comparator): In patients diagnosed with PDPH, three consecutive days of sham a-tDCS are performed starting from the day of diagnosis
  Interventions: Device: sham in therapeutic tDCS (Th-tDCS): anodal transcranial Direct Current Stimulation (a-tDCS)
- preventive a-tDCS (Pr-tDCS) (Experimental): Patients undergoing a lumbar puncture for diagnostic purposes receive an active a-tDCS intervention for three consecutive days.
  Interventions: Device: active in preventive tDCS (Pr-tDCS): anodal transcranial Direct Current Stimulation (a-tDCS)
- sham in preventive tDCS (Pr-tDCS) (Sham Comparator): Patients undergoing a lumbar puncture for diagnostic purposes receive an sham tDCS for three consecutive days.
  Interventions: Device: sham in preventive tDCS (Pr-tDCS): anodal transcranial Direct Current Stimulation (a-tDCS)

INTERVENTIONS:
Device: active in therapeutic tDCS (Th-tDCS): anodal transcranial Direct Current Stimulation (a-tDCS) — Active in therapeutic tDCS (Th-tDCS) in patients diagnosed with PDPH. The stimulations were delivered using a battery-driven direct current stimulator (HDCstim-DC stimulator, Newronika S.r.l. Milano - Italy). The current was administered through a pair of saline-soaked surface electrodes. The anode, measuring 3x3 cm, was placed over the primary motor cortex (M1) in the dominant hemisphere. This location was identified using the International 10-20 EEG system for C3 (left M1) or C4 (right M1). The cathode, measuring 6x4 cm, was positioned over the contralateral supraorbital region, immediately below the Fp position.
  In the active a-tDCS groups, each session consisted of 20 minutes stimulation with a 2 mA intensity for 3 consecutive days.
  Arms: therapeutic a-tDCS (Th-tDCS)
Device: sham in therapeutic tDCS (Th-tDCS): anodal transcranial Direct Current Stimulation (a-tDCS) — Sham in therapeutic tDCS (Th-tDCS) in patients diagnosed with PDPH. In the sham tDCS groups, the duration and electrodes application were the same of active in therapeutic tDCS (Th-tDCS), but the current was stopped 30 s thereafter. The subject felt the initial itching sensation, but no changes in cortical excitability are produced
  Arms: sham in therapeutic t-DCS (Th-tDCS)
Device: active in preventive tDCS (Pr-tDCS): anodal transcranial Direct Current Stimulation (a-tDCS) — Active in preventive tDCS (Pr-tDCS) in patients who have undergone a lumbar puncture for diagnostic purposes. The stimulations were delivered using a battery-driven direct current stimulator (HDCstim-DC stimulator, Newronika S.r.l. Milano - Italy). The current was administered through a pair of saline-soaked surface electrodes. The anode, measuring 3x3 cm, was placed over the primary motor cortex (M1) in the dominant hemisphere. This location was identified using the International 10-20 EEG system for C3 (left M1) or C4 (right M1). The cathode, measuring 6x4 cm, was positioned over the contralateral supraorbital region, immediately below the Fp position.
  In the active a-tDCS groups, each session consisted of 20 minutes stimulation with a 2 mA intensity for 3 consecutive days.
  Arms: preventive a-tDCS (Pr-tDCS)
Device: sham in preventive tDCS (Pr-tDCS): anodal transcranial Direct Current Stimulation (a-tDCS) — Sham in preventive tDCS (Pr-tDCS) in patients who have undergone a lumbar puncture for diagnostic purposes. In the sham tDCS groups, the duration and electrodes application were the same of active in preventive tDCS (Pr-tDCS), but the current was stopped 30 s thereafter. The subject felt the initial itching sensation, but no changes in cortical excitability are produced
  Arms: sham in preventive tDCS (Pr-tDCS)

SUMMARY:
Post-dural puncture headache (PDPH) is the most prevalent complication in patients undergoing diagnostic or therapeutic lumbar puncture (LP). The pathophysiology of PDPH is primarily attributed to the mechanical traction on pain-sensitive intracranial nerves (e.g., the upper cervical, 5th, 9th, and 10th cranial nerves) and vascular structures, mediated by persistent dural damage leading to cerebrospinal fluid (CSF) leakage and subsequent CSF pressure reduction.

According to the International Classification of Headache Disorders 3rd edition (ICHD3), PDPH is classified as a headache subtype due to low CSF pressure. It typically manifests as an orthostatic headache within a few days post-LP, accompanied by symptoms such as neck pain, tinnitus, auditory changes, photophobia, and nausea. While PDPH usually resolves within 7-10 days, it can result in extended hospital stays and increased need for medication. The use of atraumatic needles is the most effective preventive measure for PDPH, though other commonly recommended practices such as bed rest, fluid administration, and caffeine have questionable efficacy.

Transcranial direct current stimulation (tDCS) is a non-invasive brain stimulation (NIBS) technique that applies low-voltage electrical currents through surface electrodes on the scalp. Depending on the stimulation type-anodal or cathodal-tDCS can induce long-lasting increases or decreases in neuronal excitability and vascular-neuronal activity coupling. Research has shown that anodal tDCS (a-tDCS) applied to the primary motor cortex (M1) can alleviate various pain conditions, including fibromyalgia, neuropathic pain, and headaches. The pain-relieving effects of M1 a-tDCS are believed to follow the modulation of intracortical inhibitory GABAergic transmission, and the descending connections from M1 to the thalamus and periaqueductal gray.

Although short-term a-tDCS treatment has shown promise in preventing migraines and medication-overuse headaches, its role in preventing and treating PDPH remains unexplored. This study aims to evaluate the efficacy of preventive and therapeutic a-tDCS applied to M1 in patients undergoing diagnostic LP.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75 years;
* indication to undergo diagnostic lumbar puncture LP.

Exclusion Criteria:

* any prior exposure to brain stimulation;
* contraindications to tDCS;
* a previous diagnosis of migraine or chronic headache;
* usage of preventive medication at the baseline assessment;
* history of depression
* obesity
* multiple lumbar puncture LP attempts.
* cognitive impairment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | From enrollment to the end of treatment at 1 week
  The primary outcome was to assess differences between the two groups in PDPH-related pain, evaluated using the Visual Analogue Scale (VAS) and referred to pain intensity at that specific moment. The VAS is a self administered scale in which patients indicate the intensity of pain experienced by selecting a point on a continuous line ranging from 0 to 100 mm, representing the absence of pain to the worst pain, respectively. This scale is widely used in pain studies, with demonstrated validity and reproducibility. In the Th-tDCS study, VAS was administered at T0, before starting tDCS, and two hours before and two hours after the tDCS sessions (T1, T2, T3, T4, and T5).
  In the Pr-tDCS study, VAS was administered each day at the end of tDCS sessions (T0, T1, and T2).

SECONDARY OUTCOMES:
Brief Pain Inventory (BPI) | From enrollment to the end of treatment at one week
  As secondary outcome we analyzed the effects of tDCS on other pain-related symptoms associated with LP, evaluated using the Brief Pain Inventory (BPI). The BPI is a multidimensional measurement tool originally developed to assess the intensity and interference of pain in cancer patients. In this study, the BPI was used to assess painful symptoms associated with LP, evaluating both the intensity of pain and its interference with affective and activity aspects of the patient's daily life over the past 24 hours.
  In the Th-tDCS study, the BPI was collected before starting tDCS (T0) and two hours after the last tDCS stimulation (T5). In the Pr-tDCS study, the BPI was collected before starting tDCS (T0) and two hours after the last stimulation (T2).

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Neuromed, Pozzilli, Isernia, Italy

REFERENCES:
- [Background] Ornello R, Caponnetto V, Ratti S, D'Aurizio G, Rosignoli C, Pistoia F, Ferrara M, Sacco S, D'Atri A. Which is the best transcranial direct current stimulation protocol for migraine prevention? A systematic review and critical appraisal of randomized controlled trials. J Headache Pain. 2021 Nov 27;22(1):144. doi: 10.1186/s10194-021-01361-0. PMID 34837963
- [Background] Dasilva AF, Mendonca ME, Zaghi S, Lopes M, Dossantos MF, Spierings EL, Bajwa Z, Datta A, Bikson M, Fregni F. tDCS-induced analgesia and electrical fields in pain-related neural networks in chronic migraine. Headache. 2012 Sep;52(8):1283-95. doi: 10.1111/j.1526-4610.2012.02141.x. Epub 2012 Apr 18. PMID 22512348
- [Background] Auvichayapat P, Janyacharoen T, Rotenberg A, Tiamkao S, Krisanaprakornkit T, Sinawat S, Punjaruk W, Thinkhamrop B, Auvichayapat N. Migraine prophylaxis by anodal transcranial direct current stimulation, a randomized, placebo-controlled trial. J Med Assoc Thai. 2012 Aug;95(8):1003-12. PMID 23061303
- [Background] Cerrahoglu Sirin T, Aksu S, Hasirci Bayir BR, Ulukan C, Karamursel S, Kurt A, Baykan B. Is Allodynia a Determinant Factor in the Effectiveness of Transcranial Direct Current Stimulation in the Prophylaxis of Migraine? Neuromodulation. 2021 Jul;24(5):899-909. doi: 10.1111/ner.13409. Epub 2021 May 31. PMID 34058041
- [Background] De Icco R, Putorti A, De Paoli I, Ferrara E, Cremascoli R, Terzaghi M, Toscano G, Allena M, Martinelli D, Cosentino G, Grillo V, Colagiorgio P, Versino M, Manni R, Sances G, Sandrini G, Tassorelli C. Anodal transcranial direct current stimulation in chronic migraine and medication overuse headache: A pilot double-blind randomized sham-controlled trial. Clin Neurophysiol. 2021 Jan;132(1):126-136. doi: 10.1016/j.clinph.2020.10.014. Epub 2020 Nov 5. PMID 33271482
- [Background] Meeker TJ, Keaser ML, Khan SA, Gullapalli RP, Seminowicz DA, Greenspan JD. Non-invasive Motor Cortex Neuromodulation Reduces Secondary Hyperalgesia and Enhances Activation of the Descending Pain Modulatory Network. Front Neurosci. 2019 May 8;13:467. doi: 10.3389/fnins.2019.00467. eCollection 2019. PMID 31139047
- [Background] Naegel S, Biermann J, Theysohn N, Kleinschnitz C, Diener HC, Katsarava Z, Obermann M, Holle D. Polarity-specific modulation of pain processing by transcranial direct current stimulation - a blinded longitudinal fMRI study. J Headache Pain. 2018 Oct 24;19(1):99. doi: 10.1186/s10194-018-0924-5. PMID 30355321
- [Background] Lefaucheur JP. Pain. Handb Clin Neurol. 2013;116:423-40. doi: 10.1016/B978-0-444-53497-2.00035-8. PMID 24112914
- [Background] Fregni F, El-Hagrassy MM, Pacheco-Barrios K, Carvalho S, Leite J, Simis M, Brunelin J, Nakamura-Palacios EM, Marangolo P, Venkatasubramanian G, San-Juan D, Caumo W, Bikson M, Brunoni AR; Neuromodulation Center Working Group. Evidence-Based Guidelines and Secondary Meta-Analysis for the Use of Transcranial Direct Current Stimulation in Neurological and Psychiatric Disorders. Int J Neuropsychopharmacol. 2021 Apr 21;24(4):256-313. doi: 10.1093/ijnp/pyaa051. PMID 32710772
- [Background] Lefaucheur JP. Cortical neurostimulation for neuropathic pain: state of the art and perspectives. Pain. 2016 Feb;157 Suppl 1:S81-S89. doi: 10.1097/j.pain.0000000000000401. PMID 26785160
- [Background] Knotkova H, Hamani C, Sivanesan E, Le Beuffe MFE, Moon JY, Cohen SP, Huntoon MA. Neuromodulation for chronic pain. Lancet. 2021 May 29;397(10289):2111-2124. doi: 10.1016/S0140-6736(21)00794-7. PMID 34062145
- [Background] Nitsche MA, Fricke K, Henschke U, Schlitterlau A, Liebetanz D, Lang N, Henning S, Tergau F, Paulus W. Pharmacological modulation of cortical excitability shifts induced by transcranial direct current stimulation in humans. J Physiol. 2003 Nov 15;553(Pt 1):293-301. doi: 10.1113/jphysiol.2003.049916. Epub 2003 Aug 29. PMID 12949224
- [Background] Lefaucheur JP, Antal A, Ayache SS, Benninger DH, Brunelin J, Cogiamanian F, Cotelli M, De Ridder D, Ferrucci R, Langguth B, Marangolo P, Mylius V, Nitsche MA, Padberg F, Palm U, Poulet E, Priori A, Rossi S, Schecklmann M, Vanneste S, Ziemann U, Garcia-Larrea L, Paulus W. Evidence-based guidelines on the therapeutic use of transcranial direct current stimulation (tDCS). Clin Neurophysiol. 2017 Jan;128(1):56-92. doi: 10.1016/j.clinph.2016.10.087. Epub 2016 Oct 29. PMID 27866120
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] Arévalo-Rodríguez I, Ciapponi A, Munoz L, et al (2011) Posture and fluids for preventing post-dural puncture headache. In: Arévalo-Rodríguez I (ed) Cochrane Database of Systematic Reviews. John Wiley & Sons, Ltd, Chichester, UK
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Li H, Wang Y, Oprea AD, Li J. Postdural Puncture Headache-Risks and Current Treatment. Curr Pain Headache Rep. 2022 Jun;26(6):441-452. doi: 10.1007/s11916-022-01041-x. Epub 2022 Mar 30. PMID 35353358
- [Background] Cognat E, Koehl B, Lilamand M, Goutagny S, Belbachir A, de Charentenay L, Guiddir T, Zetlaoui P, Roos C, Paquet C. Preventing Post-Lumbar Puncture Headache. Ann Emerg Med. 2021 Sep;78(3):443-450. doi: 10.1016/j.annemergmed.2021.02.019. Epub 2021 May 7. PMID 33966935
- [Derived] Gjikolaj B, Stampanoni Bassi M, Bruno A, De Ioanni V, Dolcetti E, Peter S, Galifi G, Conte A, Gilio L, Centonze D, Buttari F. Effect of Anodal Transcranial Direct Current Stimulation on the Intensity of Post-dural Puncture Headache: Results of Two Randomized Sham Controlled Trials. Neurol Ther. 2025 Jun;14(3):989-1006. doi: 10.1007/s40120-025-00734-w. Epub 2025 Apr 22. PMID 40261600